CLINICAL TRIAL: NCT01147159
Title: Biological Standardization of Allergen Extracts of Pollens of Betula Pendula, Phleum Pratense and Mite Extract of Dermatophagoides Pteronyssinus in Patients With Rhinoconjunctivitis With/ Without Asthma Sensitized to Betula Pendula, Dermatophagoides Pteronyssinus and Phleum Pratense An Open-label, Single-center Study
Brief Title: Biological Standardization of Allergen Extracts of Pollens of Betula Pendula, Phleum Pratense and Mite Extract of Dermatophagoides Pteronyssinus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roxall Medicina España S.A (Industry)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BIA-STD-001
Record Dates: First submitted 2010-05-25; First posted 2010-06-22 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Skin prick test of extracts of allergens in 4 tenfold dilutions.

ARMS (1):
- Skin Prick Test (Other)
  Interventions: Other: Extracts of allergens

INTERVENTIONS:
Other: Extracts of allergens — Skin prick test of extracts of allergens in 4 tenfold dilutions. Assessment wheal size after 15 minutes

SUMMARY:
Allergen extracts are complex mixtures of proteins and contain varying amounts of allergenic and non-allergenic components. Many factors such as the biovariability, differences in extraction process and subsequent handling of allergens can affect the final composition, potency, and stability of allergen preparations. Genetic diversity of affected people adds another level of complexity. In order to control variability and to achieve consistency and reproducibility for optimal safety and sensitivity/specificity, it is essential to standardize the amount of allergen used in prick tests. Therefore, the system for biological standardization mainly used in Europe still is the biological calibration of in-House Reference Preparations (IHRP). The method has been adopted by the Nordic Council on Medicines as the Nordic Biological Unit, Histamine Equivalent Potency (HEP) or Skin Prick Test (SPT) value. The aim of this procedure is to estimate the biological activity of allergen extracts. The activity of an allergen extract is defined as 10,000 Diagnostic Biological Units (DBU) per ml (1 SPT per ml), when the extract provokes a specific skin reaction with a wheal of the same size as a wheal provoked by reference histamine at a concentration of 10 mg/ml, when both solutions are administrated using the same technique (prick testing) on at least 20 individuals who are clinically allergic and cutaneously reactive to the allergen concerned.

The present study aims to standardize the allergen extracts of Betula pendula, Phleum pratense and Dermatophagoides pteronyssinus by using this method.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Positive clinical history with inhalant allergy to at least one of the allergen to be standardized.
* At least one positive prick test (mean wheal diameter = 3mm) when tested with already standardized extracts of the allergens under investigation.
* Positive prick test (wheal diameter =3 mm) to Histamine 10 mg/ml
* Age: 18-60 years
* Written informed consent

Exclusion criteria:

* Diseases or medications, influencing the skin tests or that contradict the correct conduct and evaluation of the study.
* Pregnancy, skin irritations, drug and alcohol abuse and participation in another clinical trial within the last 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Wheal size area | 15 minutes after skin prick test
  The primary efficacy variable will be the wheal size area of the immediate phase reaction in mm2

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zentrum für klinische Forschung Clinical Trials Center, University Hospital and University Zurich, Zurich, Switzerland